CLINICAL TRIAL: NCT02817464
Title: A Two-part, Phase 1, Exploratory and Dose-range Finding Study to Evaluate Suppression of Ovulation and Pharmacokinetics of Medroxyprogesterone Acetate Following a Single Subcutaneous Administration of TV-46046 in Women With Ovulatory Cycle
Brief Title: Study to Evaluate Suppression of Ovulation and Pharmacokinetics of Medroxyprogesterone Acetate Following Administration of TV-46046 in Women With Ovulatory Cycle
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: TV46046-WH-10075
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-06

CONDITIONS: Pregnancy; Contraception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TV-46046 - 1 (Experimental)
  Interventions: Drug: TV-46046 - 400 mg/mL
- TV-46046 - 2 (Experimental)
  Interventions: Drug: TV-46046 - 200 mg/mL

INTERVENTIONS:
Drug: TV-46046 - 400 mg/mL — A single subcutaneous injection in the abdomen of undiluted TV-46046 - 400 mg/mL
  Arms: TV-46046 - 1
Drug: TV-46046 - 200 mg/mL — A single subcutaneous injection in the abdomen of saline-diluted TV-46046 - 200 mg/mL
  Arms: TV-46046 - 2

SUMMARY:
The purpose of this pharmacodynamic and pharmacokinetic study is to identify a dose of TV-46046 (within the range 80 to 300 mg) that is both safe and consistent with contraceptive effect when injected every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* has regular menstrual cycle (24 to 35 days)
* is at low risk of pregnancy (ie, sterilized, in exclusively same-sex partnership, in monogamous relationship with vasectomized partner, or using non-hormonal IUD)
* is in good general health as determined by a medical history and physical examination
* is not pregnant and does not have desire to become pregnant in the subsequent 36 months
* has had a normal mammogram within the last year (for Part 1 only)

  * additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* has hypertension:

  * systolic blood pressure (BP) ≥160 mm Hg or diastolic BP ≥100 mm Hg
  * vascular disease
* has current or history of ischemic heart disease
* has history of stroke
* has history of thromboembolic event
* has systemic lupus erythematosus

  * positive (or unknown) antiphospholipid antibodies
  * severe thrombocytopenia
* has rheumatoid arthritis on immunosuppressive therapy
* has migraine with aura
* has unexplained vaginal bleeding
* has diabetes
* has strong family history of breast cancer (defined as one or more first degree relatives, breast cancer occurring before menopause in three or more family members, regardless of degree of relationship, and any male family member with breast cancer), or current or history of breast cancer, or undiagnosed mass detected by breast exam
* has current or history of cervical cancer
* has severe cirrhosis (decompensated) or liver tumors
* has known significant renal disease
* used Depo-Provera Contraceptive Injection or Depo-subcutaneous Provera 104 (DMPA) products in the past 12 months
* used any of the following medications within 1 month prior to enrollment:

  * any investigational drug
  * prohibited drugs per protocol
  * oral contraceptives, contraceptive ring or patch
  * levonorgestrel intrauterine system (LNG IUS) or contraceptive implant
* used a combined injectable contraceptive in the past 6 months
* less than 3 months since the end of last pregnancy
* currently lactating
* is using or plans to use prohibited drugs per protocol in the next 18 months
* has known sensitivity to MPA or inactive ingredients
* has a plan to move to another location in the next 24 months
* in the opinion of the investigator, potentially at elevated risk of HIV infection (eg, HIV -positive partner, IV drug use by self or by partner)

  * additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (2):
- United States (2):
  - Teva Investigational Site 001, Philadelphia, Pennsylvania
  - Teva Investigational Site 002, Norfolk, Virginia

REFERENCES:
- [Derived] Halpern V, Wheeless A, Brache V, Lendvay A, Cochon L, Taylor D, Dorflinger LJ. A randomized crossover study to evaluate local tolerability following subcutaneous administration of a new depot medroxyprogesterone acetate contraceptive formulation. Contracept X. 2023 Sep 12;5:100100. doi: 10.1016/j.conx.2023.100100. eCollection 2023. PMID 37823034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part study: Part 1 (Exploratory Pharmacokinetics [PK]) and Part 2 (Dose-range Finding).
Pre-assignment Details: Due to suboptimal long-term stability and re-suspendability of the TV-46046 formulation, the decision was made not to initiate Part 2 of this clinical study, and to conduct a new dose-range finding study. Participants were planned to be assigned sequentially in 3 treatment groups in Part 1. The results of the first 2 groups did not warrant the evaluation of the intermediate concentration of TV-46046 and treatment group 3 was therefore not enrolled.
Groups:
- Group 1 (TV-46046 - Undiluted): Participants received a single subcutaneous (SC) injection of undiluted TV-46046.
- Group 2 (TV-46046 - Saline-diluted): Participants received a single SC injection of saline-diluted TV-46046.
Period: Overall Study
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Started | 6 | 6
Received at Least 1 Dose of Study Drug | 6 | 6
Completed | 4 | 5
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Discontinued early due to personal decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated population included all screened participants who were enrolled and received a dose of study drug.
Groups:
- Group 1 (TV-46046 - Undiluted): Participants received a single SC injection of undiluted TV-46046.
- Total: Total of all reporting groups
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (4.04) | 34.2 (5.08) | 31.8 (5.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Serum Medroxyprogesterone Acetate (MPA) Concentration at Day 1
Description: 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Time Frame: Day 1
Population: Primary evaluable population: a subset of treated population, excluding participants who had detectable MPA in their baseline specimen or for whom a major protocol violation occurred at enrollment, including: absence of a confirmed ovulation in pre-treatment period; body mass index (BMI) outside the eligible range; or use of drugs known to impact ovulation or pharmacokinetic (PK) of MPA (with the exception of selective cyclooxygenase-2 [COX-2] inhibitors that were taken for <5 consecutive days).
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 5
nanograms (ng)/milliliter (mL) | 0.36 (0.13) | 0.67 (0.22)

2. Primary Outcome: Part 1: Serum MPA Concentration at Day 7
Time Frame: Day 7
Population: Primary evaluable population: a subset of treated population, excluding participants who had detectable MPA in baseline specimen or for whom a major protocol violation occurred at enrollment, including: absence of a confirmed ovulation in pre-treatment period; BMI outside eligible range; or use of drugs that impact ovulation or PK of MPA (exception: selective COX-2 inhibitors taken for <5 consecutive days). Overall number of participants analyzed= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 5 | 6
ng/mL | 0.37 (0.10) | 0.70 (0.22)

3. Primary Outcome: Part 1: Serum MPA Concentration at Day 28
Time Frame: Day 28
Population: Primary evaluable population: a subset of treated population, excluding participants who had detectable MPA in baseline specimen or for whom a major protocol violation occurred at enrollment, including: absence of a confirmed ovulation in pre-treatment period; BMI outside eligible range; or use of drugs that impact ovulation or PK of MPA (exception: selective COX-2 inhibitors taken for <5 consecutive days).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 6
ng/mL | 0.36 (0.07) | 0.69 (0.25)

4. Primary Outcome: Part 1: Serum MPA Concentration at Day 91
Time Frame: Day 91
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 6
ng/mL | 0.41 (0.13) | 0.62 (0.09)

5. Primary Outcome: Part 1: Serum MPA Concentration at Day 182
Time Frame: Day 182
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 5
ng/mL | 0.22 (0.08) | 0.17 (0.10)

6. Primary Outcome: Part 1: Serum MPA Concentration at Day 210
Time Frame: Day 210
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 5 | 5
ng/mL | 0.20 (0.05) | 0.12 (0.09)

7. Primary Outcome: Part 1: Maximum Observed Serum Concentration (Cmax) of MPA
Time Frame: Day 0 up to Week 52
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 6
ng/mL | 0.53 [0.43 to 0.64] | 0.97 [0.73 to 1.29]
Statistical Analysis 1: Comparison: Group 1 (TV-46046 - Undiluted) vs Group 2 (TV-46046 - Saline-diluted); Test type: Other; Geometric Mean Ratio = 1.84, 90% CI 2-sided [1.44 to 2.36]

8. Primary Outcome: Part 1: Observed Serum Drug Concentration at Day 182 (C182) of MPA
Time Frame: Day 182
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 5
ng/mL | 0.21 [0.14 to 0.31] | 0.14 [0.05 to 0.40]
Statistical Analysis 1: Comparison: Group 1 (TV-46046 - Undiluted) vs Group 2 (TV-46046 - Saline-diluted); Test type: Other; Geometric Mean Ratio = 0.66, 90% CI 2-sided [0.33 to 1.33]

9. Primary Outcome: Part 1: Time to Reach Cmax (Tmax) of MPA
Time Frame: Day 0 up to Week 52
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 6
days | 9.49 [1.96 to 40.96] | 47.99 [7.10 to 84.01]

10. Primary Outcome: Part 1: Area Under the Serum Drug Concentration by Time Curve From Time 0 to Day 182 (AUC0-182) of MPA
Time Frame: Day 0 up to Day 182
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: days*ng/mL
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 6
days*ng/mL | 58.61 [44.75 to 76.76] | 97.72 [82.20 to 116.18]
Statistical Analysis 1: Comparison: Group 1 (TV-46046 - Undiluted) vs Group 2 (TV-46046 - Saline-diluted); Test type: Other; Geometric Mean Ratio = 1.67, 90% CI 2-sided [1.33 to 2.09]

11. Primary Outcome: Part 1: Area Under the Serum Drug Concentration by Time Curve From Time 0 to Day 210 (AUC0-210) of MPA
Time Frame: Day 0 up to Day 210
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: days*ng/mL
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 6
days*ng/mL | 63.91 [48.78 to 83.74] | 103.11 [88.40 to 120.27]
Statistical Analysis 1: Comparison: Group 1 (TV-46046 - Undiluted) vs Group 2 (TV-46046 - Saline-diluted); Test type: Other; Geometric Mean Ratio = 1.61, 90% CI 2-sided [1.30 to 2.01]

12. Primary Outcome: Part 1: Area Under the Serum Drug Concentration by Time Curve From Time 0 to Infinity (AUC0-∞) of MPA
Time Frame: Day 0 up to Week 52
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: days*ng/mL
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 6
days*ng/mL | 94.56 [81.16 to 110.16] | 114.13 [98.77 to 131.88]
Statistical Analysis 1: Comparison: Group 1 (TV-46046 - Undiluted) vs Group 2 (TV-46046 - Saline-diluted); Test type: Other; Geometric Mean Ratio = 1.21, 90% CI 2-sided [1.04 to 1.40]

13. Primary Outcome: Part 1: Apparent Terminal Half-life (t1/2) of MPA
Time Frame: Day 0 up to Week 52
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: days
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 6
days | 82.87 [32.12 to 213.80] | 42.34 [23.20 to 77.28]
Statistical Analysis 1: Comparison: Group 1 (TV-46046 - Undiluted) vs Group 2 (TV-46046 - Saline-diluted); Test type: Other; Geometric Mean Ratio = 0.51, 90% CI 2-sided [0.23 to 1.13]

14. Primary Outcome: Part 2: Time to Ovulation
Description: Ovulation was defined as a single elevated serum progesterone ≥4.7 ng/mL.
Time Frame: Day 0 up to Week 78
Population: Data for this outcome measure were not collected and analyzed as Part 2 of the study was not initiated.
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Part 1: Time to Ovulation
Description: Ovulation was defined as a single elevated serum progesterone ≥4.7 ng/mL. Time to ovulation was computed as the difference in days between detection of the first post-randomization elevated progesterone and the date of treatment initiation. Median time to ovulation was derived using Kaplan-Meier estimate.
Time Frame: Day 0 up to Week 78
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 6
days | 328 [279 to 434] | 251 [196 to 291]
Statistical Analysis 1: Comparison: Group 1 (TV-46046 - Undiluted) vs Group 2 (TV-46046 - Saline-diluted); Test type: Other; p = 0.0073, Log Rank

16. Secondary Outcome: Part 2: Cmax of MPA
Time Frame: Day 0 up to Week 52
Population: Data for this outcome measure were not collected and analyzed as Part 2 of the study was not initiated.
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Part 2: Tmax of MPA
Time Frame: Day 0 up to Week 52
Population: Data for this outcome measure were not collected and analyzed as Part 2 of the study was not initiated.
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Part 2: Observed Serum Drug Concentration at Day 210 (C210) of MPA
Time Frame: Day 0 up to Day 210
Population: Data for this outcome measure were not collected and analyzed as Part 2 of the study was not initiated.
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Part 2: C182 of MPA
Time Frame: Day 0 up to Day 182
Population: Data for this outcome measure were not collected and analyzed as Part 2 of the study was not initiated.
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Part 2: AUC0-182 of MPA
Time Frame: Day 0 up to Day 182
Population: Data for this outcome measure were not collected and analyzed as Part 2 of the study was not initiated.
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Part 2: AUC0-210 of MPA
Time Frame: Day 0 up to Day 210
Population: Data for this outcome measure were not collected and analyzed as Part 2 of the study was not initiated.
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Part 2: AUC0-∞ of MPA
Time Frame: Day 0 up to Week 52
Population: Data for this outcome measure were not collected and analyzed as Part 2 of the study was not initiated.
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Part 2: Apparent Terminal Half Life (t1/2) of MPA
Time Frame: Day 0 up to Week 52
Population: Data for this outcome measure were not collected and analyzed as Part 2 of the study was not initiated.
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. AEs were considered TEAEs if onset occurred on or after the first dose date. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Day 0 up to Week 78
Population: Treated population included all screened participants who were enrolled and received a dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
Number analyzed (Participants) | 6 | 6
Participants | 6 | 6

ADVERSE EVENTS:
Time Frame: Day 0 up to Week 78
Arm/Group | Group 1 (TV-46046 - Undiluted) | Group 2 (TV-46046 - Saline-diluted)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (TV-46046 - Undiluted) (N=6) | Group 2 (TV-46046 - Saline-diluted) (N=6)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (TV-46046 - Undiluted) (N=6) | Group 2 (TV-46046 - Saline-diluted) (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 5 (5) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Urticaria (Immune system disorders) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (3)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nose injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was planned to be conducted in 2 parts (Part 1: Exploratory PK, and Part 2: Dose-range Finding). Due to suboptimal long-term stability and re-suspendability, the decision was made not to initiate Part 2 of this clinical study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT02817464/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT02817464/SAP_001.pdf